CLINICAL TRIAL: NCT02146079
Title: A Single-centre, Parallel-group, Randomised, Double-blind, Placebocontrolled, Multiple-dose Trial to Assess the Pharmacokinetics, Pharmacodynamics, and the Safety and Tolerability of Semaglutide in Healthy Male Japanese and Caucasian Subjects
Brief Title: A Trial to Assess the Pharmacokinetics, Pharmacodynamics, and the Safety and Tolerability of Semaglutide in Healthy Male Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-3634; U1111-1147-6660 (Other: WHO); JapicCTI-142550 (Registry Identifier: JAPIC)
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Semaglutide 0.5 mg (Experimental): Dose-escalation trial
  Interventions: Drug: semaglutide
- Semaglutide placebo 0.5 mg (Placebo Comparator)
  Interventions: Drug: placebo
- Semaglutide 1.0 mg (Experimental): Dose-escalation trial
  Interventions: Drug: semaglutide
- Semaglutide placebo 1.0 mg (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Subjects will be randomised to receive either semaglutide 0.5 mg, semaglutide 0.5 mg placebo, semaglutide 1.0 mg or semaglutide 1.0 mg placebo within each group. Treatment with active drug or placebo blinded within each dose level. After randomisation, the subjects will follow a fixed dose escalation. The maintenance dose of 0.5 mg will be reached after 4 weeks of 0.25 mg. The maintenance dose of 1.0 mg will be reached after 8 weeks (4 weeks) of 0.25 mg and 4 weeks of 0.5 mg). Once-weekly subcutaneous (s.c., under the skin) administration. Trial duration per subject is 18 to 21 weeks depending on the individual subject's schedule
  Arms: Semaglutide 0.5 mg; Semaglutide 1.0 mg
Drug: placebo — Subjects will be randomised to receive either semaglutide 0.5 mg, semaglutide 0.5 mg placebo, semaglutide 1.0 mg or semaglutide 1.0 mg placebo within each group. Treatment with active drug or placebo blinded within each dose level. After randomisation, the subjects will follow a fixed dose escalation. The maintenance dose of 0.5 mg will be reached after 4 weeks of 0.25 mg. The maintenance dose of 1.0 mg will be reached after 8 weeks (4 weeks) of 0.25 mg and 4 weeks of 0.5 mg). Once-weekly subcutaneous (s.c., under the skin) administration. Trial duration per subject is 18 to 21 weeks depending on the individual subject's schedule.
  Arms: Semaglutide placebo 0.5 mg; Semaglutide placebo 1.0 mg

SUMMARY:
This trial is conducted in Asia. The aim of the trial is to investigate the pharmacokinetics (the exposure of the trial drug in the body), pharmacodynamics (the effect of the investigated drug on the body), and the safety and tolerability of semaglutide in healthy male Japanese and Caucasian subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Japanese and Caucasian subjects
* Age between 20 and 55 years (both inclusive) at the time of signing informed consent
* Body weight of equal to or above 54.0 kg
* Body mass index (BMI) between 20.0 and 25.0 kg/m^2 (both inclusive)
* Glycosylated haemoglobin A1c (HbA1c) below or equal to 6.0%
* For Japanese subjects only: both parents Japanese
* For Caucasian subjects only: both parents Caucasian

Exclusion Criteria:

* Any clinically significant disease history, in the opinion of the investigator, or systemic or organ disease including: cardiological, pulmonary, gastrointestinal, hepatic, neurologic, renal, genitourinary and endocrine, dermatologic or hematologic diseases
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2 (MEN2)
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Calcitonin above or equal to 50 ng/L
* History of alcohol abuse within 1 year from screening, or a positive result in the alcohol breath test, or consumption of more than 21 units of alcohol weekly: 1 unit of alcohol equals approximately 250 mL of beer or lager, or approximately120 mL (one glass) of wine or Japanese sake, or approximately 20 mL of spirits
* Smoking of more than 5 cigarettes (including nicotine substitute products) or the equivalent, per day or unwilling to refrain from smoking whenever required for the trial procedure
* Use of prescription drugs within 3 weeks or 5 times the half-life, whichever is longer, prior to Visit 2 (randomisation), non-prescription drugs within 1 week prior to Visit 2 (randomisation). The use of vitamins, minerals and nutritional supplements, and the occasional use of paracetamol (acetaminophen) or acetylsalicylic acid are permitted

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05-21 (Actual); Primary Completion 2014-10-20 (Actual); Study Completion 2014-10-20 (Actual)

PRIMARY OUTCOMES:
Area under the plasma semaglutide concentration-time curve | During a dosing interval (0-168 hours) at steady state

SECONDARY OUTCOMES:
Maximum observed plasma semaglutide concentration at steady state | 0-168 hours after the last dose of semaglutide (0.5 and 1.0 mg)
Change in body weight from baseline to the end of treatment | Day 1 of Visit 2 (2-21 days after Visit 1), Day 92
Number of treatment emergent adverse events (TEAEs) from baseline to follow-up | From Day 1 of Visit 2 (2-21 days after Visit 1) to Day 120-127 (Visit 23)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Ikushima I, Jensen L, Flint A, Nishida T, Zacho J, Irie S. A Randomized Trial Investigating the Pharmacokinetics, Pharmacodynamics, and Safety of Subcutaneous Semaglutide Once-Weekly in Healthy Male Japanese and Caucasian Subjects. Adv Ther. 2018 Apr;35(4):531-544. doi: 10.1007/s12325-018-0677-1. Epub 2018 Mar 13. PMID 29536338
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com